CLINICAL TRIAL: NCT01956097
Title: Effects of HX106 on Improvement in Cognitive-Bio-Markers of Memory Function in Healthy Adults With Subjective Memory Complaints
Brief Title: Effects of HX106 on Improvement in Cognitive-Bio-Markers of Memory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX106
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults With Subjective Memory Complaints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HX106 590mg (Experimental): HX106 590mg/day
  Interventions: Dietary Supplement: HX106 590mg
- HX106 1180mg (Experimental): HX106 1180mg/day
  Interventions: Dietary Supplement: HX106 1180mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HX106 590mg
  Arms: HX106 590mg
Dietary Supplement: HX106 1180mg
  Arms: HX106 1180mg
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The objectives of the current study are to evaluate the efficacy and safety of HX106 in healthy adults with subjective memory complaints for improving cognitive and neurobiolgoical markers of memory.

DETAILED DESCRIPTION:
The objectives of the current study are to evaluate the efficacy and safety of HX106 in healthy adults with subjective memory complaints for improving neurocognitive functions and to find the changes of brain using magnetic resonance imaging and their associations with the neurocognitive function enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years old,
* Global Deterioration Scale score (GDS) of 2
* One or more symptoms of subjective memory impairment
* High school or higher levels of education.

Exclusion Criteria:

* Current pregnancy or breast-feeding
* Evidence of neurologic or medical conditions
* Axis I diagnosis when assessed by the board certified psychiatrist using the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV)(SCID-IV),
* One or more major depressive episode during last 12 months
* Mini-mental status examination score of 24 or less
* Clinical Dementia Rating score of 0.5 or more suggesting cognitive impairment beyond self-perceived subjective deficits
* Intelligence quotient less than 80
* Any history of head trauma involving loss of consciousness or seizure
* Contraindications to magnetic resonance imaging (MRI)
* Use of psychotropics in last 3 months
* Use of oral contraceptive medication
* Participation in other clinical trials during the study period that might affect the outcome of the present study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha W. University
Locations (1):
- Ewha W. University, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- HX106 590mg: HX106 590mg/day
  HX106 590mg
- HX106 1180mg: HX106 1180mg/day
  HX106 1180mg
Period: Overall Study
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Started | 30 | 30 | 15
Completed | 24 | 28 | 15
Not Completed | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HX106 590mg | HX106 1180mg | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 15 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 15 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.7) | 42.5 (11.2) | 40.6 (12.7) | 40.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 4 | 39
  Male | 12 | 13 | 11 | 36
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 15 | 75

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Working Memory Domain Z-score
Description: To assess the working memory performance, four well-established tests, including the symbol span from the Wechsler Memory Scale-IV, immediate recall domain from the Rey-Osterrieth Complex Figure Test, digit span, and letter number sequencing from the Korean version of the Wechsler Adult Intelligence Scale were chosen.
  Each test score was adjusted with age, sex, intelligent quotient, years of education, and baseline test scores. The adjusted test scores were then standardized into z-scores using all participants' means and standard deviations. The relative improvement (positive z-scores) or decline (negative z-scores) in performance was measured in a unit-free manner using the obtained z-scores. The individual z-scores of each test were averaged to the composite score for working memory domain.
Time Frame: Baseline, 8th week
Measure: Mean (Standard Error); unit: z-score
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Number analyzed (Participants) | 30 | 30 | 15
z-score
  baseline | -0.21955 (0.04450) | -0.15432 (0.03883) | -0.08842 (0.06861)
  week8 | 0.29594 (0.16938) | 0.34061 (0.13436) | -0.27524 (0.13489)

2. Primary Outcome: Changes From Baseline in White Matter Integrity Assessment
Time Frame: Baseline, 8th weeks
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 1st week
Population: 2 participants in the "HX106 590mg" group and 1 participant in the "HX106 1180mg" were dropped out.
Measure: Number; unit: number of participants
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Number analyzed (Participants) | 28 | 29 | 15
number of participants | 17 | 13 | 0

4. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 4th weeks
Population: 3 participants in the "HX106 590mg" group and 1 participant in the "HX106 1180mg" were dropped out.
Measure: Number; unit: number of participants
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Number analyzed (Participants) | 27 | 29 | 15
number of participants | 16 | 18 | 7

5. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: 8th weeks
Population: 6 participants in the "HX106 590mg" group and 2 participant in the "HX106 1180mg" were dropped out.
Measure: Number; unit: number of participants
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Number analyzed (Participants) | 24 | 28 | 15
number of participants | 12 | 10 | 8

ADVERSE EVENTS:
Arm/Group | HX106 590mg | HX106 1180mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 23/30 | 22/30 | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HX106 590mg (N=30) | HX106 1180mg (N=30) | Placebo (N=15)
Autonomic symptoms: palpitations/tachycardia (Cardiac disorders) | 3 | 2 | 1 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: accomodation disturbances (Eye disorders) | 3 | 0 | 2 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: diarrhea (Gastrointestinal disorders) | 1 | 0 | 2 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: constipation (Gastrointestinal disorders) | 4 | 2 | 0 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: nausea/vomitting (Gastrointestinal disorders) | 2 | 2 | 2 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: weight gain (General disorders) | 6 | 3 | 0 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: weight loss (General disorders) | 4 | 0 | 2 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: headache (General disorders) | 6 | 6 | 5 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: orthostatic dizziness (General disorders) | 5 | 2 | 2 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: increased tendency to sweating (General disorders) | 2 | 1 | 2 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: reduced salivation (General disorders) | 0 | 1 | 1 — any of the side effects listed in the UKU side effect rating scale
Neurologic symptoms: dystonia (Nervous system disorders) | 0 | 1 | 2 — any of the side effects listed in the UKU side effect rating scale
Neurologic symptoms: rigidity (Nervous system disorders) | 2 | 2 | 2 — any of the side effects listed in the UKU side effect rating scale
Neurologic symptoms: paresthesia (Nervous system disorders) | 3 | 0 | 2 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: increased fatigability (Psychiatric disorders) | 11 | 5 | 4 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: sleepiness/sedation (Psychiatric disorders) | 9 | 3 | 2 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: failing memory (Psychiatric disorders) | 3 | 1 | 1 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: depression (Psychiatric disorders) | 4 | 1 | 3 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: tension/inner unrest (Psychiatric disorders) | 0 | 1 | 2 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: increased duration of sleep (Psychiatric disorders) | 2 | 2 | 1 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: reduced duration of sleep (Psychiatric disorders) | 7 | 2 | 1 — any of the side effects listed in the UKU side effect rating scale
Psychic symptoms: increased dream activity (Psychiatric disorders) | 5 | 2 | 1 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: micturition disturbances (Renal and urinary disorders) | 0 | 0 | 1 — any of the side effects listed in the UKU side effect rating scale
Autonomic symptoms: polyuria/polydipsia (Renal and urinary disorders) | 1 | 4 | 1 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: increased sexual desire (Reproductive system and breast disorders) | 0 | 0 | 1 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: morbilliform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: cannot be classified (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — any of the side effects listed in the UKU side effect rating scale
Other symptoms: pruritus (Skin and subcutaneous tissue disorders) | 4 | 7 | 2 — any of the side effects listed in the UKU side effect rating scale

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No